CLINICAL TRIAL: NCT04499833
Title: Evaluation of the HepatoPredict Prognostic Tool in the Decision of Liver Transplant in Hepatocellular Carcinoma
Brief Title: HepatoPredict Prognostic Tool for the Decision of Liver Transplant in Hepatocellular Carcinoma
Acronym: HepatoPredict
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Collaborators: Ophiomics - Precision Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHULC.CI.HCC.2020
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma, Scirrhous; Recurrence Tumor
Keywords: cirrhosis; Hepatocellular Carcinoma; liver transplant; tumor recurrence; biomarkers; prognosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence; Fibrosis | interventions — Liver Transplantation

STUDY DESIGN:
Intervention Model Description: Prospective evaluation of patients with hepatocellular carcinoma in cirrhotic liver, outside the "Milan Criteria" for liver transplant, that comply with the morphologic criteria stablished for the proposed HepatoPredict Tool: (1) Total tumour volume below 500 cm3; (2) Total number of tumour lesions below 10; and (3) maximum individual tumour diameter below 10 cm. Those patients are proposed to be submitted to molecular study of the hepatocellular carcinoma and, if comply with the "HepatoPredict genomic signature", liver transplantation will be proposed. Patients will be followed up for up to 5 years after transplantation for survival and survival-free-of-disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- liver transplant outside the "Milan Criteria" (Experimental): patients with hepatocellular carcinoma, outside the "Milan Criteria", that complied with the proposed HepatoPredictTool, submitted to liver transplant
  Interventions: Procedure: liver transplant

INTERVENTIONS:
Procedure: liver transplant — liver transplant

SUMMARY:
Liver transplant is the most effective treatment for hepatocellular carcinoma (HCC) in cirrhosis. Due to organs shortage, the proper selection of patients is imperative. Prevailing clinical morphological models used in most centres (Milan Criteria), can exclude potential candidates and include patients with aggressive biological behaviour. To more accurately select candidates for liver transplant, the inclusion of criteria that could predict the behaviour and aggressiveness of tumours, such as molecular markers, might be useful.

The investigators propose the use of a new algorithm (HepatoPredict Prognostic Tool), that combine clinical and molecular criteria that address the biology of tumours, in a single centre prospective, intervention study. Data from the "HepatoPredict genomic signature" are added to the clinical and imagiology algorithm. Based on this tool, patients outside the usual eligibility criteria for liver transplant will be proposed for this treatment. These patients will be transplanted with marginal livers or with livers from patients with Familial Amyloid Polyneuropathy, not competing with patients on the waiting list. Patients will be followed up to 60 months after transplant, to assess survival and HCC recurrence with biannual imagiology screening. Survival and disease-free-survival rates will be compared with those obtained by the usual management of patients included and excluded by Milan Criteria.

DETAILED DESCRIPTION:
Liver transplant is the most effective treatment for hepatocellular carcinoma (HCC) in cirrhosis. Due to organs shortage, the proper selection of patients is imperative. Prevailing clinical morphological models used in most centres (Milan Criteria), can exclude potential candidates and include patients with aggressive biological behaviour. To more accurately select candidates for liver transplant, the inclusion of criteria that could predict the behaviour and aggressiveness of tumours, such as molecular markers, might be useful. The investigators propose the use of a new algorithm (HepatoPredict Prognostic Tool, Ophiomics), combining morphologic information, clinical and molecular criteria, in a prospective, intervention, single centre study.

Patients aged 18 to 70 years, with HCC in cirrhosis, not eligible for liver transplant under the "Milan Criteria", whom had the following morphologic characteristics: total tumour volume below 500 cm3, total number of tumour lesions below 10 and maximum individual tumour diameter below 10 cm, will be proposed for the "HepatoPredict genomic signature" analysis (Ophiomics), obtained from DNA of tumor samples. Those considered candidates by the algorithm are to be proposed for transplant with marginal livers or with livers from patients with Familial Amyloid Polyneuropathy.

Patients will be followed up to 60 months after transplant, to assess survival and HCC recurrence with biannual imagiology screening by triphasic CT scan. Additionally, circulating tumour DNA will be assessed previously to the transplant and biannually for up to 60 months. Survival and disease-free-survival rates will be compared with those obtained with the usual management of patients included and excluded by Milan Criteria, both in the same referral transplant center and in the published literature.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma associated with cirrhosis
* Ages between 18 and 70 years
* Total tumour volume below 500 cm3
* Total number of tumour lesions below 10
* Maximum individual tumour diameter below 10 cm

Exclusion Criteria:

* eligible under the "Milan Criteria"

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
death | from 6 months after liver transplant up to 60 months
  death by any cause
hepatocellular carcinoma recurrence | from 6 months after liver transplant up to 60 months
  identification of hepatocellular carcinoma recurrence through biannual triphasic CT scan

SECONDARY OUTCOMES:
hepatocellular carcinoma recurrence through liquid biopsy | from 6 months after liver transplant up to 60 months
  early identification of hepatocellular carcinoma DNA through biannual serum samples (liquid biopsy)

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Pinto-Marques, MD PhD, Principal Investigator — Centro Hospitalar Universitário de Lisboa Central
Locations (1):
- Centro Hepato-bilio-pancreático e de Transplantação do Hospital Curry Cabral, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No